CLINICAL TRIAL: NCT05222321
Title: Sensory-Play Based (SenPlay) Intervention for Young Children With or At Risk for Attention Deficit Hyper Activity Disorder (ADHD)
Brief Title: Sensory-Play Based (SenPlay) Intervention for Young Children With or At Risk for ADHD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed by the IRB when PI did not submit for annual review.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14128
Record Dates: First submitted 2022-01-18; First posted 2022-02-03 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention; Focused attention; Sensory; Play-based intervention; Occupational therapy; Pediatrics
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methods

STUDY DESIGN:
Intervention Model Description: To address the aims of this study, the investigators will recruit 20 participants and utilize a randomized, experimental study with a two-group longitudinal, pre-posttest, linear association study design to measure attention levels and off-task behaviors. This is the first step in determining the effects of the SenPlay intervention on focused attention. The intervention will occur over three time points in a clinic therapy room and occupational therapy gym in an outpatient pediatric clinic.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be aware of group assignment, but will be notified of their group assignment at the end of the three intervention sessions upon request. The percentage of on and off-task behaviors will be calculated by two coders, blinded to the group assignment will code session. Prior to the study, both coders will achieve a reliability of at least 95% accuracy in training sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SenPlay Intervention Group (Experimental): SenPlay is a sensory-play based intervention that includes deep tactile pressure, vestibular and proprioceptive input as a therapeutic medium to facilitate optimal arousal through activities such as pushing, pulling, climbing, jumping, and crashing. These activities are designed to facilitate changes in the child's arousal by providing sensory input and are used at random during the 15 minute window and are facilitated and monitored to ensure the child is reaching a threshold of moderate to vigorous physical activity. All participants will wear the ActiGraph accelerometer to measure the intensity of physical activity during the SenPlay intervention. Intervention sessions will occur at three time points, one per week for three weeks. Following the SenPlay intervention, participants will engage in 10 minutes of developmentally appropriate tasks (DAT) lead by the same investigator. DAT will be videotaped and coded for off task behaviors using Momentary Time Sampling (MTS).
  Interventions: Other: Sensory-Play Based (SenPlay) Intervention
- Free play Control Group (Placebo Comparator): The control group will engage in spontaneous, free play with the investigator supervising only for safety within the sensorimotor gym for 15 minutes, prior to the assessment of off-task behaviors during 10 minutes of developmentally appropriate tasks (DAT). All participants will wear the ActiGraph accelerometer to measure the intensity of physical activity reached during spontaneous, free play. Participants in the control group will participate in three sessions, one per week for three weeks. Intervention sessions will occur at three time points, one per week for three weeks. Following the spontaneous play, participants will engage in 10 minutes of developmentally appropriate tasks (DAT) lead by the same investigator. DAT will be videotaped and coded for off task behaviors using Momentary Time Sampling (MTS).
  Interventions: Other: Spontaneous, Free Play

INTERVENTIONS:
Other: Sensory-Play Based (SenPlay) Intervention — SenPlay is a sensory-play based intervention that includes deep tactile pressure, vestibular and proprioceptive input as a therapeutic medium to facilitate optimal arousal through sensory-play based activities such as pushing, pulling, climbing, jumping, crashing, and swinging. These activities are designed to facilitate changes in the child's arousal through providing sensory input to ensure the child is reaching a threshold of moderate to vigorous physical activity. Completed at three time points, once weekly for three weeks.
  Arms: SenPlay Intervention Group
Other: Spontaneous, Free Play — Participant engages in spontaneous, free play with the investigator supervising only for safety within the sensorimotor gym for 15 minutes. Completed at three time points, once weekly for three weeks.
  Arms: Free play Control Group

SUMMARY:
The purpose of this pilot study is to determine the effects of 15 minutes of sensory-play based (SenPlay) intervention on improving focused attention in developmentally appropriate tasks in young children with or at risk for ADHD.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, written consent will be obtained by the investigators. Twenty participants will be recruited for this randomized, experimental study with a two-group longitudinal, pre-posttest, linear association study design to measure attention levels and off-task behaviors. All participants will attend a total of four sessions. The investigator, a registered, licensed occupational therapist, will lead all intervention sessions utilizing a set protocol. Participants will complete an intake session to determine baseline fine motor skills for developmentally appropriate tasks (DAT) before being randomly assigned to either the control group or the SenPlay intervention group. The control group will engage in spontaneous, free play with the supervising only for safety within the sensorimotor gym (see image 1) for 15 minutes, prior to the assessment of off-task behaviors during 10 minutes of DAT. The intervention group will engage in 15-minutes of SenPlay intervention, followed by assessment of off-task behaviors during 10 minutes of DAT. The 10 minutes of DAT will be coded at the beginning of each 15 second interval (Wood et al., 2016) for a total of 40 observation periods. The percentage of on and off-task behaviors will be calculated. Two coders, blinded to the group assignment will code session. Prior to the study, both coders will achieve a reliability of at least 95% accuracy in training sessions.

ELIGIBILITY:
Inclusion Criteria

* Age 3-years, to 5-years, 11-months
* Diagnosis or provisional diagnosis of ADHD or overactivity by the primary care physician, psychologist or neurologist
* No diagnosis of neurological disorders other than ADHD
* Normal or corrected vision
* Cognitive skills to follow verbal instruction
* Gross and fine motor skills to engage in sensorimotor activities and school readiness tasks

Exclusion Criteria:

* Participants will be excluded if they currently take medication for ADHD or exhibit severe physical impairments that result in inability to engage in the SenPlay intervention, fine motor and visual motor activities.

Ages: 36 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Change in focused attention as measured by Momentary Time Sampling from intervention one to intervention three. | Intervention session one (week one) to intervention session three (week three).
  Momentary Time Sampling (MTS) using a MTS observation chart will be used to code on and off task behaviors when engaged in developmentally appropriate task (DAT) for three sessions per participant. Sessions will be recorded using a video camera and coded to ensure completeness of data tracking for on and off-task behaviors. Using MTS, the child's behavior is coded at the beginning of every 15 second time interval using a stopwatch to ensure 15 second intervals. Focused attention will be measured by calculating the percentage of on and off-task behaviors with all data collection and coding methods being the same for all participants in both groups. On-task behaviors are operational defined as behaviors in which both the eyes and hands are focused on the task, appropriately responding to the investigator's verbal instruction, and manipulation of materials as instructed by the investigator while off-task behaviors include any behavior not meeting the criteria of an on-task behavior.

SECONDARY OUTCOMES:
Intensity of physical activity measured at all intervention sessions | Three time points, once weekly for three weeks.
  The ActiGraph (GTX3) accelerometer will be used to measure the intensity of physical activity (PA) for each child while engaged in the SenPlay intervention and spontaneous, free play.

CONTACTS AND LOCATIONS:
Overall Officials: Thubi Kolobe, PT, Ph.D., Principal Investigator — University of Oklahoma
Locations (1):
- Sensational Kids, Inc, Yukon, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
No identifiable study data will be shared with any outside entities. The subject's information will not be used or distributed for future research studies even if identifiers are removed.

REFERENCES:
- [Result] Acar IH, Frohn S, Prokasky A, Molfese VJ, Bates JE. Examining the Associations Between Performance Based and Ratings of Focused Attention in Toddlers: Are We Measuring the Same Constructs? Infant Child Dev. 2019 Jan-Feb;28(1):e2116. doi: 10.1002/icd.2116. Epub 2018 Oct 22. PMID 30853857
- [Result] Barton EE, Reichow B, Schnitz A, Smith IC, Sherlock D. A systematic review of sensory-based treatments for children with disabilities. Res Dev Disabil. 2015 Feb;37:64-80. doi: 10.1016/j.ridd.2014.11.006. Epub 2014 Nov 25. PMID 25460221
- [Result] Gaertner BM, Spinrad TL, Eisenberg N. Focused Attention in Toddlers: Measurement, Stability, and Relations to Negative Emotion and Parenting. Infant Child Dev. 2008 Aug;17(4):339-363. doi: 10.1002/ICD.580. PMID 19112517
- [Result] Lin CL, Min YF, Chou LW, Lin CK. Effectiveness of sensory processing strategies on activity level in inclusive preschool classrooms. Neuropsychiatr Dis Treat. 2012;8:475-81. doi: 10.2147/NDT.S37146. Epub 2012 Oct 23. PMID 23118541
- [Result] Mangeot SD, Miller LJ, McIntosh DN, McGrath-Clarke J, Simon J, Hagerman RJ, Goldson E. Sensory modulation dysfunction in children with attention-deficit-hyperactivity disorder. Dev Med Child Neurol. 2001 Jun;43(6):399-406. doi: 10.1017/s0012162201000743. PMID 11409829
- [Result] Miller LJ, Coll JR, Schoen SA. A randomized controlled pilot study of the effectiveness of occupational therapy for children with sensory modulation disorder. Am J Occup Ther. 2007 Mar-Apr;61(2):228-38. doi: 10.5014/ajot.61.2.228. PMID 17436845
- [Result] Miller LJ, Nielsen DM, Schoen SA. Attention deficit hyperactivity disorder and sensory modulation disorder: a comparison of behavior and physiology. Res Dev Disabil. 2012 May-Jun;33(3):804-18. doi: 10.1016/j.ridd.2011.12.005. Epub 2012 Jan 11. PMID 22236629
- [Result] NICHD Early Child Care Research Network. Predicting individual differences in attention, memory, and planning in first graders from experiences at home, child care, and school. Dev Psychol. 2005 Jan;41(1):99-114. doi: 10.1037/0012-1649.41.1.99. PMID 15656741
- [Result] Wan Yunus F, Liu KP, Bissett M, Penkala S. Sensory-Based Intervention for Children with Behavioral Problems: A Systematic Review. J Autism Dev Disord. 2015 Nov;45(11):3565-79. doi: 10.1007/s10803-015-2503-9. PMID 26092640
- [Result] Zentall SS, Zentall TR. Optimal stimulation: a model of disordered activity and performance in normal and deviant children. Psychol Bull. 1983 Nov;94(3):446-71. No abstract available. PMID 6657825
- [Result] Fedewa AL, Erwin HE. Stability balls and students with attention and hyperactivity concerns: implications for on-task and in-seat behavior. Am J Occup Ther. 2011 Jul-Aug;65(4):393-9. doi: 10.5014/ajot.2011.000554. PMID 21834454
- [Result] Mah, J, Doherty, M. Sensorimotor intervention group for children with ADHD and sensory processing difficulties: A feasibility study. Journal of Child and Family Studies. 2021; 30, 447-459.
- [Result] McGoey, K. Schreiber, J, Venesky, L., Westwood, W., McGuirk, L., Schaffner, K. Factor structure of attention deficit hyperactivity disorder symptoms for children age 3 to 5 years. Journal of Psychoeducational Assessment. 2015; 33(5), 430-438
- [Result] Olson LJ, Moulton HJ. Use of weighted vests in pediatric occupational therapy practice. Phys Occup Ther Pediatr. 2004;24(3):45-60. doi: 10.1300/j006v24n03_04. PMID 15257968
- [Result] Pollock, N. Sensory integration: A review of the current state of the evidence, Occupational Therapy Now. 2009; 11
- [Result] Posner MI, Rothbart MK. Research on attention networks as a model for the integration of psychological science. Annu Rev Psychol. 2007;58:1-23. doi: 10.1146/annurev.psych.58.110405.085516. PMID 17029565
- [Result] Schilling DL, Washington K, Billingsley FF, Deitz J. Classroom seating for children with attention deficit hyperactivity disorder: therapy balls versus chairs. Am J Occup Ther. 2003 Sep-Oct;57(5):534-41. doi: 10.5014/ajot.57.5.534. PMID 14527115
- [Result] Seifert, AM. Metz, AE. The effects of inflated seating cushions on engagement in preschool circle time. Early Childhood Education Journal. 2016; 45(3), 411-418
- [Result] Sirard, J., Trost, S., Pfeiffer, K., Dowda, M., Pate, R. Calibration and evaluation of an objective measure of physical activity in preschool children. Journal of Physical Activity and Health. 2005; 3, 345-357
- [Result] Wood, BK., Hojnoski, RL., Laracy, SD., Olson, CL. Comparison of observational methods and their relation to ratings of engagement in young children. Topics in Early Childhood Special Education. 2016; 35, 211-222
- [Result] Zakszeski, BN., Hojnoski, RL., Wood, BK. Considerations for Time Sampling Interval Durations in the Measurement of Young Children's Classroom Engagement. Topics in Early Childhood Special Education. 2017; 37(1), 42-53